CLINICAL TRIAL: NCT00665938
Title: Followup of Infants Fed Non-routine Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Kim Merkel, Mead Johnson
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 3369-6; 3369-6
Record Dates: First submitted 2008-03-28; First posted 2008-04-24 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Physical development
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator)
  Interventions: Other: Infant formula
- 2 (Experimental)
  Interventions: Other: Infant formula
- 3 (Experimental)
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Infant formula — Arm 1. extensively hydrolyzed infant formula without probiotics (Nutramigen LIPIL)
  Arm 2. partially hydrolyzed infant formula with probiotics
  Arm 3. extensively hydrolyzed infant formula with probiotics
  Other Names: No other names are applicable to the 3 intervention arms

SUMMARY:
The purpose of this study is to compare physical development of infants fed one of three study formulas.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study 3369-5

Exclusion Criteria:

* None

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Estimated)
Dates: Start 2006-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Achieved weight | 5 years

SECONDARY OUTCOMES:
Tolerance | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Deolinda Scalabrin, MD, Study Director — Mead Johnson Nutrition